CLINICAL TRIAL: NCT00586183
Title: Cardiac Sympathetic Activity in Patients With the Apical Ballooning Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Abhiram Prasad, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 06-002093
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2006-03

CONDITIONS: Apical Ballooning Syndrome
Keywords: Ventricular Remodeling
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Ventricular Remodeling | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The subject will then be positioned in the PET scanner . After optimal positioning of the left ventricle within the field of view, a transmission scan will be performed with either a germanium-68 or CT source for subsequent attenuation correction.
  Interventions: Procedure: PET scan

INTERVENTIONS:
Procedure: PET scan — The subject will then be positioned in the PET scanner . After optimal positioning of the left ventricle within the field of view, a transmission scan will be performed with either a germanium-68 or CT source for subsequent attenuation correction.
  Other Names: Positron emission scan

SUMMARY:
Our hypothesis is that altered cardiac sympathetic activity is present and may contribute to the myocardial stunning observed in the apical ballooning syndrome.

Aim: Assess the extent and reversibility of cardiac adrenergic neuronal dysfunction using carbon-11 hydroxyephedrine (C-11 HED), a positron emission tomography (PET) tracer, in patients with the apical ballooning syndrome.

DETAILED DESCRIPTION:
General methods: Five patients will undergo PET scans within a few days of or during the initial hospital admission for apical ballooning syndrome and during follow-up at 4 to 6 weeks to evaluate regional perfusion using N-13 ammonia and cardiac sympathetic activity with C-11 HED.

PET scanning protocol On the morning of the study, patients will arrive at the Mayo Clinic PET Imaging Center in a fasting state. The use of medications will be ascertained and recorded. An intravenous cannula will be placed in each arm. The subject will then be positioned in the PET scanner . After optimal positioning of the left ventricle within the field of view, a transmission scan will be performed with either a germanium-68 or CT source for subsequent attenuation correction. The PET scanning sequence is outlined below. Because 11C-HED uptake is dependent on flow characteristics, a flow study will be performed using N-13 ammonia. N-13 ammonia (10 to 20 mCi) will be injected over 20 seconds, and dynamic acquisition will be performed for 20 minutes with the following sequence:16 frames at 3 seconds, 10 frames at 12 seconds, and 2 frames at 240 seconds. Following a 50-minute period of N-13 ammonia decay, 11C-HED (20mCi) will be injected over 30 seconds, and a dynamic acquisition will be performed with the following sequence: 6 frames at 30 seconds, 2 frames at 60 seconds, 2 frames at 150 seconds, 2 frames at 300 seconds, 2 frames at 600 seconds, and 1 frames at 1,200 seconds. To correct for 11C-metabolites in the blood activity, venous samples will be drawn at 0, 1, 5, 10, 20, 40, and 60 minutes (total ~25 ml of blood) after the injection of C-11 HED. Heart rate, systemic blood pressure, and a 12-lead electrocardiogram will be obtained noninvasively with each peak isotope activity.

ELIGIBILITY:
Inclusion Criteria:

* Transient akinesis or dyskinesis of the left ventricular apical and mid-ventricular segments with regional wall-motion abnormalities extending beyond a single epicardial vascular distribution.
* Absence of obstructive coronary disease or angiographic evidence of acute plaque rupture.
* New electrocardiographic abnormalities (either ST-segment elevation or T-wave inversion.
* Absence of recent significant head trauma, intracranial bleeding, pheochromocytoma, myocarditis, hypertrophic cardiomyopathy.

Exclusion Criteria:

* Hemodynamically unstable patients (requiring pressor support) will be excluded.
* Breastfeeding women.
* Pregnant women (urine pregnancy test required within 48 hours prior to each set of PET scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Assess the extent and reversibility of cardiac adrenergic neuronal dysfunction | During PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Abhiram Prasad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States